CLINICAL TRIAL: NCT05947942
Title: Thoracic Fluid Content by Electrical Cardiometry Versus Diaphragmatic Excursion by Ultrasound for Prediction of Weaning Success in Patients With Lung Congestion
Brief Title: Thoracic Fluid Content for Weaning Parameters
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Shawky Elshaer, Doctor, Benha University
Other Study IDs: MD.10.4.2023
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Lung; Congestive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to compare the thoracic fluid content measured by electrical cardiometry versus the diaphragmatic excursion measured by ultrasound for prediction of weaning success in patients having lung congestion.

DETAILED DESCRIPTION:
lung congestion was defined as distention of blood vessels in the lungs and filling of the alveoli with fluid as a result of an infection, high blood pressure, or cardiac insufficiencies (i.e., inability of the heart to function adequately.

The process of weaning from ventilatory support takes almost 40% of the time spent on ventilator. Weaning indices like spontaneous tidal volumes, minute ventilation and rapid shallow breathing index, have been used extensively in clinical practice for weaning purposes . These parameters measure the overall respiratory volumes produced by the muscles of breathing and do not take into account the independent contribution of the diaphragm. During resting, the main muscle of breathing is the diaphragm .

Diaphragmatic excursion is the movement of the thoracic diaphragm during breathing. Normal diaphragmatic excursion should be 3-5 cm, but can be increased in well-conditioned persons to 7-8 cm. This measures the contraction of the diaphragm. Diaphragmatic excursion is positively correlated with lung inspiratory volumes and can accurately reflect the muscle strength and function . Diaphragmatic excursion is an index for respiratory muscle fatigue during the spontaneous breathing trial (SBT).

Thoracic fluid content (TFC) is one of the many variables measured by the ICON electrical cardiometry (EC) device. The ICON device is one relatively new proprietary implementation of impedance cardiography technology, which is also often called thoracic electrical bioimpedance .

Impedance cardiography is based on measuring the changes in total resistance of the thorax to electric current. The impedance to electric current is determined by the resistance of different tissues such as bone, muscles, and fluids. The fluid compartment is considered the dynamic component that would cause short term changes in thoracic impedance . TFC is calculated as the reciprocal of the total thoracic impedance and is considered a numerical measure of total (intravascular and extravascular) thoracic fluid . Although TFC is a measure of both extra and intravascular thoracic fluid, it might provide an estimate of the increase in intrathoracic fluids such as to facilitate the risk of pulmonary congestion , we hypothesized that TFC, as an estimate of lung congestion, can serve as predictor for weaning outcomes in critically ill patient.

ELIGIBILITY:
Inclusion Criteria:

* • Patients of both genders aged 18-70 years old.

  * Acute Physiology and Chronic Health Evaluation II (APACHE II) score
  * Patients with congested lung including; Acute exacerbation of COPD patients with acute respiratory failure (PaO2/FiO2 ratio ≤300 or PaCO2 ≥ 50 mm Hg at intubation), pneumonia, chronic kidney disease, heart failure (New York Heart Association Classification III, IV) who will be candidate for weaning from invasive mechanical ventilation according to the treating physician's judgement using the ICU weaning protocol.

Exclusion Criteria:

* • Patients younger than 18 years or older than 70 years

  * Refusal to participate.
  * Obesity (BMI≥35).
  * Pregnancy.
  * Patients with pneumothorax, pleural, or pericardial effusion, lung contusion, and thoracotomy.
  * Hepatic dysfunction.
  * history or new detection of paralysis (no movement) or paradoxical movement of a single hemidiaphragm.
  * preexisting cervical spinal injury, history of neuromuscular disorders
  * Patients with injuries, burns, or wounds which precluded the proper application of the device electrodes will be also excluded from the study.
  * Mechanical ventilation < 48 hrs

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on 100 patients admitted to critical care department at Benha university hospitals with lung congestion. Patients who are candidate for weaning from invasive mechanical ventilation (after 48 h) and who agree to participate in the study will be involved.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-03-20 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Thoracic fluid content by electrical cardiometry versus diaphragmatic excursion by Ultrasound for prediction of weaning success in patients with lung congestion | 1 year
  compare the thoracic fluid content measured by electrical cardiometry versus the diaphragmatic excursion measured by ultrasound for prediction of weaning success in patients having lung congestion.

CONTACTS AND LOCATIONS:
Locations (1):
- Shawky meselhi shawky, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No